CLINICAL TRIAL: NCT03657602
Title: Immediate Postpartum Insertion of Kyleena vs Mirena Contraceptive Intrauterine Devices
Brief Title: Immediate Postpartum Insertion of Contraceptive Intrauterine Devices
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9588
Record Dates: First submitted 2018-08-24; First posted 2018-09-05 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated one to one to the Kyleena or Mirena group and assessment will occur in parallel
Who Masked: Participant
Masking Description: Participant will be blinded to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Contraceptive Kyleena (Experimental): Determination of expulsion and discontinuation rates in participants randomly allocated to receive levonorgestrel intrauterine systems Kyleena Intrauterine System
  Interventions: Drug: Kyleena Intrauterine System
- Contraceptive Mirena (Experimental): Determination of expulsion and discontinuation rates in participants randomly allocated to receive levonorgestrel intrauterine systems Mirena Intrauterine System
  Interventions: Drug: Mirena Intrauterine System

INTERVENTIONS:
Drug: Kyleena Intrauterine System — Participant will be randomly allocated to this intervention
  Other Names: levonorgestrel intrauterine system
  Arms: Contraceptive Kyleena
Drug: Mirena Intrauterine System — Participant will be randomly allocated to this intervention
  Other Names: levonorgestrel intrauterine system
  Arms: Contraceptive Mirena

SUMMARY:
In this randomized trial, investigators intend to determine the expulsion and discontinuation rate of immediate postpartum intrauterine devices in the patient population of the University of Oklahoma Women's Healthcare Specialists Clinic (OUWHSC).

DETAILED DESCRIPTION:
Between 40-57% of women report having unprotected intercourse prior to the 6 week postpartum visit. Immediate postpartum long-acting reversible contraception (LARC) is extremely important in preventing short-interval and unintended pregnancies. The postpartum period is an excellent time for intrauterine device (IUD) or implant insertion as women are often highly motivated to prevent unwanted pregnancies at this time. Per the American College of Obstetrics and Gynecology (ACOG), expulsion rates for immediate postpartum IUD insertion are higher than for interval or post-abortion insertion. Despite the higher expulsion rate of immediate postpartum IUD placement over interval placement, cost-benefit analysis data strongly suggest the superiority of immediate placement in reduction of unintended pregnancy, especially for women at greatest risk of not attending the postpartum follow-up visit. This study will randomly allocate participants one to one to the Kyleena or the Mirena IUD group, and participants will be blinded to allocation of groups. Participants will follow up at routine postpartum visit within 4 weeks of delivery, and a second follow up will be performed at 10 weeks. Ultimately, this study will attempt to provide more detailed information on the difference of rates of expulsion and discontinuation of the different-sized Mirena and Kyleena intrauterine devices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* desire an intrauterine device as postpartum contraception
* want to avoid pregnancy for at least 1 year
* are currently pregnant
* desire immediate postpartum IUD insertion.

Exclusion Criteria:

* known uterine or cervical anomaly
* untreated cervical infection
* untreated cervical infection
* pelvic infection within 3 months of the study
* recent (within last 3 months) or active intrauterine infection
* genital bleeding of unknown etiology
* history of postpartum or postabortal sepsis
* cervical cancer or carcinoma in suit
* plan to leave Tulsa area within 10 weeks postpartum
* allergy to device ingredients

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Expulsion of intrauterine contraception | within 10 weeks of placement
  IUD string check and ultrasound check

SECONDARY OUTCOMES:
Discontinuation of intrauterine contraception | Through study completion, an average of 1 year
  Date IUD is removed

CONTACTS AND LOCATIONS:
Overall Officials: Valorie Owens, MSW, Study Director — University of Oklahoma
Locations (1):
- University of Oklahoma - Tulsa, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No